CLINICAL TRIAL: NCT02216851
Title: A Randomized, Open Label, No-treatment Controlled, Multi-center, Efficacy and Safety Study Using Restylane Perlane to Shape the Nasal Dorsum and/or Nasal Root
Brief Title: Restylane Perlane to Shape the Nasal Dorsum and/or Nasal Root
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH1310
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Results first posted 2021-09-23 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2021-09

CONDITIONS: Nasal Augmentation
Keywords: hyaluronic acid; no-treatment control; enhancement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restylane Perlane (Experimental): Single injection of Restylane Perlane in nasal dorsum and/or nasal root
  Interventions: Device: Restylane Perlane
- No-treatment control (No Intervention): No-treatment control group do not receive any treatment during the main study period

INTERVENTIONS:
Device: Restylane Perlane — Intradermal injection
  Arms: Restylane Perlane

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using Restylane Perlane to shape the nasal dorsum and/or nasal root in comparison with a no-treatment control group

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin
* Subject with desire to shape the nasal dorsum and/or nasal root
* Subjects who, in the opinion of the investigator, can achieve a clinically meaningful aesthetic correction of their nose with ≤ 1 ml Restylane Perlane

Exclusion Criteria:

* Subjects with previous nasal surgery, including grafts or implants to the nose area
* Subjects requiring filler treatment around the tip of the nose or between the eyebrows (glabella region) to achieve a good aesthetic outcome
* Subjects with a history of chronic sinusitis or rhinitis
* Subjects who have previously received aesthetic treatment in the forehead, glabellar and/or nose area with a dermal filler

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q-Med AB, Study Director — Galderma R&D
Locations (2):
- China (2):
  - Beijing
  - Guangzhou

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Perlane | No-treatment Control
Started | 98 | 33
Completed | 96 | 32
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Perlane | No-treatment Control | Total
Number analyzed (Participants) | 98 | 33 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 33 | 131
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 33 | 127
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 98 | 33 | 131
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference of Change in Volume (mL) at 6 Months After Baseline Versus Pre-treatment in the Nasal Dorsum/Nasal Root Between Restylane Perlane Treatment Group and No-treatment Control
Description: The primary objective of the study was to evaluate the efficacy of Restylane Perlane in shaping the nasal dorsum and/or nasal root as compared to no-treatment control, by assessment of the primary endpoint:The change in volume will be measured using 3 D photography technique.
  The change in volume was calculated as the value at 6 months of treatment group compared with non-treatment group
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mL
Arm/Group | Restylane Perlane | No-treatment Control
Number analyzed (Participants) | 98 | 33
mL | 0.82 (0.03) | 0.11 (0.03)

ADVERSE EVENTS:
Time Frame: During study participation, up to 12 months.
Description: Each subject was questioned about AEs at each clinical visit starting at the treatment visit, Visit 2. The question asked was "Since your last clinical visit have you had any health problems?" Information on AEs could also be obtained from signs and symptoms detected during each examination, observations by the study personnel, reactions recorded in the subject diary that were ongoing on Day 14 or spontaneous reports from the subjects during the study.
Arm/Group | Restylane Perlane | No-treatment Control
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/33
Serious Adverse Events (participants affected / at risk) | 4/98 | 1/33
Other Adverse Events (participants affected / at risk) | 0/98 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restylane Perlane (N=98) | No-treatment Control (N=33)
mixed hemorrhoids (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Solid pseudopapillary tumor of the pancreas (Hepatobiliary disorders) | 1 (1) | 0 (0)
Fallopian tube obstruction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
peritoneal adhesions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes